CLINICAL TRIAL: NCT00100672
Title: Phase I Study of an Easy-to-Use Intravenous Formulation of Liposome Entrapped C-raf Antisense Oligonucleotide (LErafAON-ETU) Administered on a Weekly Schedule in Patients With Advanced Cancer
Brief Title: Study to Determine the Maximum Tolerated Dose of LErafAON in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LErafAON-ETU-104-R02
Record Dates: First submitted 2005-01-04; First posted 2005-01-05 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-06

CONDITIONS: Neoplasms
Keywords: LErafAON-ETU; Signal transduction; Neoplasm; Cancer; NeoPharm; Liposomes; Antisense; Anti-cancer; Advanced neoplasm; Advanced cancer; Chemotherapy; Refractory cancer; Metastatic cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

INTERVENTIONS:
Drug: LErafAON-ETU

SUMMARY:
The primary purpose of this study is to identify a dose of Liposome Entrapped c-raf Antisense Oligonucleotide Easy-to-Use (LErafAON-ETU) which maximizes potential benefits of the compound to patients with advanced cancer, without compromising their safety. This study will also assess the processing of LErafAON-ETU by the body over time. Patients will receive an intravenous infusion of LErafAON-ETU each week. Multiple blood samples will be taken for pharmacokinetic analysis during the first treatment; two samples will be taken during both the second and third treatments. Patients will be eligible to continue treatment until the occurrence of unacceptable toxicity or disease progression.

In LErafAON-ETU, antisense oligonucleotides specific to c-raf, are associated with liposomes, which are microscopic membrane-like structures created from lipids (fats). Raf-1 is a protein which plays a critical role in many aspects of cellular activation and growth. Therefore, it is thought to be an important factor that may support tumor development. LErafAON-ETU potentially limits the ability of a cell to produce the Raf-1 protein.

DETAILED DESCRIPTION:
This Phase I, open-label, dose-escalation study is designed to determine the maximum tolerated dose of LErafAON-ETU in patients who have advanced cancer considered unresponsive to available, conventional modalities or treatments. LErafAON-ETU will be administered as an IV infusion once weekly for 3 consecutive weeks (a Treatment Cycle). A complete pharmacokinetic profile of raf-1 antisense oligonucleotide will be assessed in week 1 only; limited pharmacokinetic sampling will be done prior to and at the end of infusion in weeks 2 and 3 only. Tumor/disease evaluation will be performed upon completion of 6 infusions (2 Cycles). Dose escalation will not occur until the safety and tolerability at a given dose level has been confirmed for 1 Cycle.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, patients must meet the following criteria:

* Be ≥18 years of age.
* Have advanced (local and/or metastatic) histologically documented cancer not considered responsive to available conventional modalities or treatment (i.e., no life prolonging therapy or therapy with a greater potential for patient benefit is available).
* Have an ECOG Performance status of 0-1.
* Have a life expectancy of >12 weeks.
* Have recovered from acute toxicities of prior treatment: *No treatment with radiotherapy or with cytotoxic or biologic agents within 3 weeks prior to study entry. At least 2 weeks must have elapsed since any prior surgery or granulocyte-stimulating growth factor therapy. Chronic treatment with non-investigational gonadotropin-releasing hormone agonists or other hormonal or supportive care is permitted. Concurrent bisphosphonate treatment is permitted if initiated ≥90 days prior to study entry. *Chronic Grade 1 toxicities due to prior treatment or other causes are permitted.
* Be in adequate condition as evidenced by the following clinical laboratory values:

  * Absolute neutrophil count (ANC) ≥1,500/mm³,
  * Hemoglobin ≥9.0 g/dL,
  * Platelets ≥125,000/mm³,
  * PT, aPTT, creatinine, calcium, and total bilirubin ≤the institutional upper limit of normal (ULN),
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x ULN,
  * Alkaline phosphatase ≤2.5 x ULN
* Patients (male and female) must be willing to practice an effective method of birth control during the study.
* Patient must understand the investigational nature of this study and sign an Institutional Review Board (IRB) approved informed consent form prior to the performance of any study specific procedure.

Exclusion Criteria:

Patients are excluded from this study for the following:

* Active uncontrolled bleeding or bleeding diathesis (e.g., active peptic ulcer disease).
* Any active infection requiring parenteral or oral antibiotic treatment.
* Known infection with human immunodeficiency virus or hepatitis virus.
* Active heart disease including myocardial infarction within the previous 6 months, symptomatic coronary artery disease, arrhythmias currently requiring medication, or congestive heart failure.
* Known or suspected active central nervous system metastasis (patients stable 8 weeks after completion of treatment for central nervous system metastasis are eligible).
* Requiring immediate palliative treatment of any kind, including surgery and/or radiotherapy
* Concurrent anti-tumor therapy (except for chronic hormonal anti-tumor therapy).
* Treatment with any investigational drug within the 30-day period prior to enrollment in the study.
* Known hypersensitivity to any of the components of LErafAON-ETU.
* Prior treatment with LErafAON (previous sonicated formulation).
* Female patients who are pregnant or breast-feeding.
* Unwilling or unable to follow protocol requirements.
* Any consideration which in the Investigator's opinion deems the patient an unsuitable candidate to receive study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-12; Primary Completion 2009-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of LErafAON-ETU.

SECONDARY OUTCOMES:
To determine the pharmacokinetics of raf antisense oligonucleotide after intravenous administration of LErafAON-ETU
To determine any anti-tumor effects of LErafAON-ETU.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - premiere Oncology-Arizona, Scottsdale, Arizona
  - Premiere Oncology-Santa Monica, Santa Monica, California